CLINICAL TRIAL: NCT01871753
Title: The Bacteriuria in Renal Transplantation (BiRT) Study: A Prospective, Randomized, Parallel-group, Multicenter, Open-label, Superiority Trial Comparing Antibiotics Versus no Treatment in the Prevention of Symptomatic Urinary Tract Infection in Kidney Transplant Recipients With Asymptomatic Bacteriuria
Brief Title: The Bacteriuria in Renal Transplantation (BiRT) Study: A Trial Comparing Antibiotics Versus no Treatment in the Prevention of Symptomatic Urinary Tract Infection in Kidney Transplant Recipients With Asymptomatic Bacteriuria
Acronym: BiRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: University Hospital, Lille (Other); Universitair Ziekenhuis Brussel (Other); Hôpital Necker Enfants-Malades, Université de Paris Descartes, APHP, France (Unknown); Centre Hospitalier Universitaire Brugmann (Other); Centre Hospitalier Universitaire de Charleroi (Other); University Ghent (Other); Centre Hospitalier Epicura, Belgium (Unknown); University of Liege (Other); Nantes University Hospital (Other)
Responsible Party: Principal Investigator, Julien Coussement, MD, Julien Coussement, MD, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BiRT study; 2012-003857-26 (EudraCT Number)
Record Dates: First submitted 2013-05-31; First posted 2013-06-07 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Asymptomatic Bacteriuria; Bacteriuria; Urinary Tract Infections; Kidney Transplantation
MeSH Terms: conditions — Bacteriuria; Urinary Tract Infections | interventions — Anti-Infective Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotics (Experimental): 10 days of antibiotics, started and selected according to the antibiogram results. In case of reinfection or relapse, re-administration of antimicrobial agents will be performed according to the antibiogram results (for a maximum of 3 cycles of ten days of antibiotics during the 12 months of the follow-up).
  Interventions: Other: Anti-Infective Agents
- No treatment (No Intervention): no antibiotics delivered in case of asymptomatic bacteriuria, independently of the number of asymptomatic episodes.

INTERVENTIONS:
Other: Anti-Infective Agents — 10 days of antibiotics, started and selected according to the antibiogram results. In case of reinfection or relapse, re-administration of antimicrobial agents will be performed according to the antibiogram results (for a maximum of 3 cycles of ten days of antibiotics during the 12 months of the follow-up)
  Other Names: Anti-Infective Agents: not applicable - no specific agent; The choice of antimicrobial agent is at the discretion of the physician, and is based on the antibiogram results
  Arms: Antibiotics

SUMMARY:
The purpose of this study is to compare antibiotics versus no-treatment in kidney transplant recipients with asymptomatic bacteriuria.

DETAILED DESCRIPTION:
The BiRT trial investigators would be interested to collaborate with some additional hospitals, particularly centers having high level of antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient with asymptomatic bacteriuria after the first two months post-transplantation

Exclusion Criteria:

* Pregnant women or women who wish to become pregnant during the course of the study
* Presence of indwelling urinary devices such as urethral catheter, ureteral catheter, nephrostomy and/or suprapubic catheter
* Combined transplantation (liver-kidney, lung-kidney, heart-kidney)
* Urinary tract surgery during the last two months
* Surgical urological procedure planned in the next 2 weeks
* Neutropenia (≤ 500 neutrophils/mm3)
* Important intensification of immunosuppression (Solumedrol bolus and/or use of thymoglobulin) or any other treatment of an acute graft rejection in the last two months
* Use of antibiotics at the time of the asymptomatic bacteriuria (except for prevention of Pneumocystis jirovecii)
* End-Stage Renal Disease (ESRD) requiring dialysis
* Non-functioning native bladder (e.g. bladder dysfunction requiring intermittent self-catheterization, orthotopic ileal neobladder)
* Recurrent acute graft pyelonephritis (≥ 2 episodes in the last year)
* Kidney transplant recipients who could not return for regular follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of a first episode of symptomatic urinary tract infection | 12 months

SECONDARY OUTCOMES:
incidence of a first episode of pyelonephritis | 12 months
clearance of asymptomatic bacteriuria | 12 months
occurrence of new episodes of asymptomatic bacteriuria | 12 months
graft function/graft survival | 12 months
incidence of graft rejection | 12 months
patient survival | 12 months
utility of a control urine culture for diagnosis of asymptomatic bacteriuria in kidney transplant recipients | 12 months
level of antimicrobial resistance in bacteria responsible for symptomatic urinary tract infections | 12 months
total number of days of antimicrobial therapy | 12 months
cost of antimicrobial treatment for asymptomatic bacteriuria and symptomatic urinary tract infection | 12 months
number of hospitalizations for asymptomatic bacteriuria and symptomatic urinary tract infection treatment | 12 months
total number of symptomatic urinary tract infections in both groups | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julien Coussement, MD, Study Director — Hôpital Universitaire Erasme, Brussels, Belgium
Locations (15):
- Belgium (8):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Centre Hospitalier Epicura, Baudour
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Hôpital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Vrije Universiteit Brussel, Brussels
  - Centre Hospitalier Universitaire de Charleroi, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Universitaire de Liège, Liège
- France (7):
  - Groupe Henri Mondor-Albert Chenevier, Assistance Publique-Hôpitaux de Paris, Créteil
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Department of Kidney Transplantation, Hôpital Necker Enfants-Malades, Université de Paris Descartes, APHP, Paris
  - Hôpital Tenon, Assistance Publique-Hôpitaux de Paris, Paris
  - Centre Hospitalier Universitaire de Saint-Étienne, Saint-Etienne
  - Centre Hospitalier Universitaire Rangueil, Toulouse